CLINICAL TRIAL: NCT04083833
Title: A Phase 1, Single Ascending Dose, Randomized, Double-Blind, Placebo and Positive Controlled Study to Evaluate the Cardiovascular Effect of Tetrodotoxin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TTX-TQT-101
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: TQT Study
Keywords: TQT TTX Halneuron cardiac safety
MeSH Terms: interventions — Tetrodotoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): (Period 1) A single TTX dose of 15 μg (0.5 mL of TTX 30 μg/mL injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet) (Period 2) A single TTX dose of 30 μg (1 mL of TTX 30 μg/mL injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet) (Period 3) A single TTX dose of 45 μg (1.5 mL of TTX 30 μg/mL injection solution) administered as 2 SC injections with a single oral moxifloxacin matching placebo (1 x placebo tablet)
  Interventions: Drug: Tetrodotoxin
- Control (Placebo Comparator): Treatment D:
  (Period 1)A single matching-TTX placebo administered with a single oral moxifloxacin matching placebo
  Treatment E:
  (Period 2)A single matching-TTX placebo with a single oral 400 mg moxifloxacin
  Treatment F:
  (Period 3)A single matching-TTX placebo with a single oral moxifloxacin matching placebo
  Treatment G:
  (Period 1)A single matching-TTX placebo with a single oral 400 mg moxifloxacin
  Treatment H:
  (Period 2)A single matching-TTX placebo with a single oral moxifloxacin matching placebo
  Treatment I:
  (Period 3)A single matching-TTX placebo with a single oral 400 mg moxifloxacin
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tetrodotoxin — A single TTX dose in a dose ascending study
  Other Names: Halneuron
  Arms: Treatment Arm
Drug: Placebos — matching placebo comparator
  Arms: Control

SUMMARY:
To determine if a single subcutaneous (SC) administration of TTX at various dose levels has an effect on the QT/QTc intervals when assessing concentration QT (C-QT) relationship (i.e., QT/QTc intervals prolongation in relation to plasma levels of TTX) in healthy adult subjects.

Secondary:

1. To determine if a single SC administration of TTX at various dose levels has an effect on other important electrocardiogram (ECG) parameters in healthy adult subjects.
2. To demonstrate sensitivity of this QTc assay using moxifloxacin as a positive control.
3. To confirm plasma pharmacokinetic (PK) of a single SC administration of TTX at various dose levels when administered to healthy adult subjects.
4. To determine the overall safety and tolerability of a single SC administration of TTX at various dose levels when administered to healthy adult subjects.

Test Product, Dose, Duration, Mode of Administration, and Batch Number:

The test product was 30 µg/mL tetrodotoxin (TTX) for injection, Lot No. F141124-001.

Subjects were also administered:

* Tetrodotoxin matching placebo a sterile 0.9% sodium chloride injection or normal saline for injection, Lot No. 84-093-DK
* 400 mg Avelox® (moxifloxacin hydrochloride) tablets, Lot No. BXHJ1S1
* Moxifloxacin matching placebo film-coated tablets, Id.-No.: K15372, Batch No.: C1606007

Treatments were as follows:

Treatment Arm (n = 9)

Treatment A:

(Period 1) A single TTX dose of 15 μg (0.5 mL of TTX 30 μg/mL injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Treatment B:

(Period 2) A single TTX dose of 30 μg (1 mL of TTX 30 μg/mL injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Treatment C:

(Period 3) A single TTX dose of 45 μg (1.5 mL of TTX 30 μg/mL injection solution) administered as 2 SC injections with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Subjects randomized to the Control Arm were further randomized to receive 1 of 2 treatment sequences (Treatment Sequence DEF [n = 8] and Treatment Sequence GHI [n = 8]):

Control Arm (n = 16)

Treatment D:

(Period 1) A single matching-TTX placebo (0.5 mL of placebo injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Treatment E:

(Period 2) A single matching-TTX placebo (1 mL of placebo injection solution) administered as 1 SC injection with a single oral 400 mg moxifloxacin (1 x 400 mg tablet)

Treatment F:

(Period 3) A single matching-TTX placebo (1.5 mL of placebo injection solution) administered as 2 SC injections with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Treatment G:

(Period 1) A single matching-TTX placebo (0.5 mL of placebo injection solution) administered as 1 SC injection with a single oral 400 mg moxifloxacin (1 x 400 mg tablet)

Treatment H:

(Period 2) A single matching-TTX placebo (1 mL of placebo injection solution) administered as 1 SC injection with a single oral moxifloxacin matching placebo (1 x placebo tablet)

Treatment I:

(Period 3) A single matching-TTX placebo (1.5 mL of placebo injection solution) administered as 2 SC injections with a single oral 400 mg moxifloxacin (1 x 400 mg tablet) All oral study drugs were administered with approximately 240 mL of water.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female 18 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose and throughout the study.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, neurologic examinations, laboratory profiles, vital signs, or ECGs, as deemed by the PI or designee.
5. For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

   * non-hormone releasing intrauterine device for at least 3 months prior to the first dose and throughout the study.
   * surgical sterilization of the partner (vasectomy for 4 months minimum prior to the first dose).
   * physical barrier method (e.g., condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study.

   A female subject who claims to be sexually inactive, but becomes sexually active during the course of the study must agree to use a physical barrier method (e.g., condom, diaphragm) with spermicide from the time of the start of sexual activity and throughout the study.

   In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 28 days following the last dose.
6. For a female of non childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
7. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose of study drug. A male who has been vasectomized less than 4 months prior to study first dose must follow the same restrictions as a non vasectomized male).
8. If male, must agree not to donate sperm from the first dose until 90 days after last dosing.
9. No clinically significant history or presence of ECG findings as judged by the PI at screening and check-in of Period 1, including each criterion as listed below:

   * Normal sinus rhythm (heart rate between 50 bpm and 100 bpm inclusive);
   * QTcF interval ≤ 450 msec;
   * QRS interval ≤ 110 msec; if > 110 msec, result will be confirmed by a manual over read;
   * PR interval ≤ 220 msec.
10. Normal renal function (creatinine clearance from 80 to 180 mL/minute per Cockcroft-Gault equation; 24-hour urinary creatinine collection may be used for borderline cases).
11. PEF of ≥ 80% per handheld meter and oxygen saturation of ≥ 95% by pulse oximetry.
12. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
5. History or presence of:

   * risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   * sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities.
6. Any acute or chronic pain conditions requiring ongoing treatment or limiting daily activities.
7. History of fainting upon blood sampling or needle puncture.
8. Findings during the screening neurological examination that could interfere with or preclude neurological assessments during the study, in the opinion of the PI or designee.
9. History or presence of neurologic or neuromuscular disease.
10. Allergy to band aids, adhesive dressing or medical tape.
11. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s), related compounds, or fish.
12. History of anaphylaxis to a medication, dietary item, or environment exposures (including bee stings).
13. Female subjects with a positive pregnancy test or lactating.
14. Positive urine drug, cotinine, or alcohol results at screening or check in of Period 1.
15. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
16. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
17. Seated heart rate is lower than 50 bpm or higher than 99 bpm at screening.
18. Unable to refrain from or anticipates the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study.
19. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dose and throughout the study.
20. Donation of blood or significant blood loss within 56 days prior to the first dose.
21. Plasma donation within 7 days prior to the first dose.
22. Participation in another clinical study within 30 days prior to the first dose. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
Cardiodynamic | 24 hours
  The primary cardiodynamic endpoint was the effect of TTX plasma concentrations on the QTc interval using linear mixed-effect exposure-response modeling, including the predicted ddQTc at Cmax values corresponding to exposure levels of interest.

SECONDARY OUTCOMES:
ECG Paramenters | 24 hours
  Other ECG parameters such as QTc, QT, PR, and RR intervals, QRS duration, and HR
ECG Paramenters | 24 hours
  Abnormalities in T wave morphology and pathologic U waves will be reported when identified by the cardiologist reviewer, as appropriate.
Assay Sensitivity | 24 hours
  3. Assay sensitivity assessment with ddQTc at the geometric mean Cmax value predicted from a linear mixed-effect model evaluating the relationship between QTc and moxifloxacin plasma concentrations (exposure-response modeling).

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No